CLINICAL TRIAL: NCT04953884
Title: Clinical Study to Investigate the Efficacy, Pharmacokinetics, Immunogenicity and Safety of Wilate in Severe Von Willebrand Disease Patients Under the Age of 6 Years
Brief Title: Efficacy, PK, Immunogenicity and Safety of Wilate in Severe Von Willebrand Disease VWD) Patients <6 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIL-33
Record Dates: First submitted 2021-06-18; First posted 2021-07-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — von Willebrand Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- wilate treatment (Experimental): PK: Single dose of 80 IU/kg body weight (BW). Prophylactic treatment: 30-50 IU/kg BW administered 2-3 times per week at the recommended dose of over 12 months. Minor haemorrhage: loading dose 30-50 IU/kg BW followed by a maintenance dose of 30-40 IU/kg BW every 12-24 hours to achieve von Willebrand factor activity (VWF:Ac) and FVIII:C trough levels of >30%. Major haemorrhage: loading dose 50-80 IU/kg BW followed by a maintenance dose of 30-50 IU/kg BW every 12-24 hours to achieve VWF:Ac and FVIII:C trough levels of >50%. Minor surgery: loading dose of 40-60 IU/kg BW followed by a maintenance dose of 20-30 IU/kg BW every 12- 24 hours for up to 3 days, to achieve VWF:Ac peak levels of 50% after loading dose and trough levels >30% during maintenance. Major surgery: loading dose of 60-80 IU/kg BW followed by a maintenance dose of 30-40 IU/kg BW every 12-24 hours for up to 6 days or longer, to achieve VWF:Ac peak levels of 100% after loading dose and trough levels >50% during maintenance
  Interventions: Drug: wilate

INTERVENTIONS:
Drug: wilate — wilate is a plasma-derived, stable, highly purified, double virus inactivated concentrate of freeze-dried active VWF and factor VIII (FVIII) prepared from cryoprecipitate and intended for the treatment of patients with von Willebrand disease (VWD) and/or haemophilia A

SUMMARY:
The WIL-33 study aims to determine the efficacy, pharmacokinetics, immunogenicity and safety of wilate as routine prophylaxis in up to 12 paediatric patients (eight evaluable) with severe von Willebrand Disease VWD (defined as screening von Willebrand factor ristocetin cofactor activity [VWF:RCo] <20%) under the age of 6 years, over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged <6 years at the time of screening
2. Type 3 (at least four patients), severe type 2 (except 2N) or severe type 1 VWD (any of which with VWF:RCo <20%) according to medical history, requiring substitution therapy with a VWF-containing product
3. Minimum body weight 12.5 kg at the time of screening
4. Voluntarily given, fully informed written and signed consent obtained before any study-related procedures are conducted (obtained from the patient's parent(s)/ legal guardian(s))

Exclusion Criteria:

1. History or current suspicion of VWF or FVIII inhibitors
2. Injection of DDAVP or VWF-containing product within 72 hours prior to inclusion
3. Medical history of a thromboembolic event
4. Platelet count <100,000/µL at screening (except for VWD type 2B)
5. Patients receiving, or scheduled to receive, immunosuppressant drugs (other than antiretroviral chemotherapy), such as prednisone (equivalent to >10 mg/day), or similar drugs
6. Treatment with any investigational medicinal product (IMP) in another interventional clinical study currently or within four weeks before enrolment
7. Other coagulation disorders or bleeding disorders
8. Known hypersensitivity to any of the components of the study drug

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Total annualised bleeding rate (tABR) during prophylactic treatment with wilate. | Up to 12 months of treatment

SECONDARY OUTCOMES:
Area under the curve (AUC) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
AUC normalised for the administered dose (AUCnorm) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
In vivo half-life (T1/2) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
Maximum plasma concentration (Cmax) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
Time to reach maximum plasma concentration (Tmax) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
Mean residence time (MRT) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
Volume of distribution (Vd) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
Clearance (CL) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline, 15 minutes, 3, 9, 24, 48 and 72 hours after dosing of 80 IU/kg BW wilate
Incremental in-vivo recovery (IVR) of wilate for VWF:Ac (VWF:RCo) and FVIII:C (OS) over time | At baseline and at 1, 2, 3, 6, 9, and 12 months of treatment
Efficacy of wilate in the prevention and treatment of spontaneous and traumatic breakthrough BEs based on their rate and the proportion of spontaneous and traumatic BEs successfully treated with wilate | Up to 12 months of treatment
  Assessed by the use of a 4-point ordinal haemostatic efficacy scale (excellent - good - moderate - none)
The overall efficacy of wilate in perioperative prophylaxis against excessive bleeding as assessed at the end of the postoperative period by the responsible treating investigator | Up to 12 months of treatment
  Assessed by the use of a 4-point ordinal haemostatic efficacy scale (excellent - good - moderate - none)
wilate consumption data for prophylactic treatment, for on-demand treatment and during surgical prophylaxis | Up to 12 months of treatment
Incidence of VWF and FVIII inhibitors | Up to 12 months of treatment
Incidence of thromboembolic events | Up to 12 months of treatment
Joint Health Status determination by the use of the Hemophilia Joint Health Score, given the patient's age and constitutional development allow this assessment | At baseline and at 12 months of treatment
Safety and tolerability of wilate assessed by monitoring adverse events (AEs) throughout the study | Up to 12 months of treatment

CONTACTS AND LOCATIONS:
Locations (9):
- Tulane University, New Orleans, Louisiana, United States
- Czechia (2):
  - University Hospital Ostrava Department for Pediatric Medicine, Ostrava
  - University Hospital Motol, Department of Paediatric Haematology and Oncology, Prague
- Gerinnungszentrum Rhein-Ruhr Ambulanz und Fachlaboratorium für Gerinnungserkrankungen/Hämophilie, Duisburg, Germany
- IMSP Mother and Child Institute, Chisinau, Moldova
- PHI University Clinic for Child Diseases, Skopje, North Macedonia
- Russia (2):
  - FSBI National Research Medical Center of Pediatric Hematology, Oncology and Immunology, Moscow
  - Morozovskaya Children's Hospital, Moscow
- Danylo Halytsky Lviv National Medical University, Communal Institution of Lviv Regional Council "Western Ukrainian Specialized Children's Medical Centre", Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No